CLINICAL TRIAL: NCT03762954
Title: Assessment of Cognitive and Functional Impairment of Older Patients After Endoscopic Retrograde Cholangiopancreatography (ERCP) and Endoscopic Ultrasound
Brief Title: Assessment of Cognitive and Functional Impairment in Older Patients After ERCP
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Patrick Yachimski, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 181485
Record Dates: First submitted 2018-11-27; First posted 2018-12-04 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Research Subjects: All adults aged 60 years or older scheduled to undergo outpatient ERCP and/or EUS at Vanderbilt University Medical Center (VUMC) will be invited to participate in the study. Invited patients who consent to participate as study subjects will undergo neurocognitive and functional assessment pre-procedure and at 90 days post-procedure.
  Interventions: Other: Neurocognitive function assessment

INTERVENTIONS:
Other: Neurocognitive function assessment — Neurocognitive function will be assessed via a phone battery derived from standard cognitive tests proven feasible and valid to assess memory, attention, reasoning, and executive functioning. Functional status will also be assessed via phone. The duration of time required for the patient to complete telephone interview for neurocognitive and functional assessment will be approximately 45 minutes per time point.

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an interventional endoscopy procedure utilized in the therapeutic management of pancreatobiliary diseases including gallstones, bile duct strictures, leaks and infections, pancreatitis, and cancers of the bile duct or pancreas. ERCP is classified as a high risk procedure. Potential adverse events directly attributable to the technical aspects of ERCP include pancreatitis, hemorrhage, infection, and bowel wall perforation. Other potential adverse events of ERCP may be less apparent and/or unknown, such as risk of neurocognitive dysfunction. Overall, neurocognitive dysfunction after medical procedures impacts quality of life, functional disability, depression, and caregiver and societal burden.

The prevalence of postoperative neurocognitive dysfunction and disability following interventional endoscopy procedures such as ERCP has not been reported. This prospective observational study is designed to assess the prevalence of cognitive impairment and functional disability after ERCP and endoscopic ultrasound (EUS) procedures in older patients, and to assess whether specific patient and/or procedural factors are associated with increased risk of adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years or older
* Scheduled to undergo outpatient ERCP and/or EUS at Vanderbilt University Medical Center (VUMC)

Exclusion Criteria:

* Age <60 years
* Inpatient status at the time of ERCP/EUS
* Documented history of dementia
* Inability to provide informed consent for study participation, implying baseline neurocognitive dysfunction
* Blind, deaf, or unable to speak English, as these conditions would preclude our ability to perform assessments.
* No access to a telephone to permit pre-procedure and 3 month post-procedure neurocognitive assessment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults aged 60 years or older scheduled to undergo outpatient ERCP and/or EUS at Vanderbilt University Medical Center (VUMC).
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of cognitive impairment and/or functional disability | 90 days
  Number of subjects with an increase in impairment and/or disability after undergoing outpatient endoscopic retrograde cholangiopancreatography (ECRP) and/or endoscopic ultrasound (EUS)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yachimski, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No